CLINICAL TRIAL: NCT02448407
Title: Intraarticular Injections of Platelet-rich Plasma in Pain's Treatment of the Osteoarthritic Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMH-PRP-2013; 2013-001303-36 (EudraCT Number)
Record Dates: First submitted 2015-04-27; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Platelet-rich plasma; Pain's treatment
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Platelet rich plasma (Experimental): Three intraarticular injection, one each fifteen days
  Interventions: Biological: Platelet rich plasma
- Hyaluronic acid (Active Comparator): Infiltrations of Hyaluronic acid as Hyaluronate 2,5 ml, 1 % solution, administered by intraarticular injection (3 doses, one each fifteen days)
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Biological: Platelet rich plasma — Three intraarticular injections of platelet-rich plasma, one each fifteen days
  Other Names: PRP, Platelet Concentrate
  Arms: Platelet rich plasma
Drug: Hyaluronic acid — Infiltrations of Hyaluronic acid as Hyaluronate 2,5 ml, 1% solution, administered by intraarticular injections (three doses, one each fifteen days)
  Other Names: Adant
  Arms: Hyaluronic acid

SUMMARY:
Platelet-rich plasma (PRP), due to its high content of cytokines, bioactive proteins and platelet growth factors, may contribute to diminish the pain of arthritic knee. It was also recently recognized a regenerative cell potential improving the concentration of hyaluronic acid and stabilizing angiogenesis in arthritic knees

This study therefore seeks to assess the analgesic power of PRP in osteoarthritic knees intraarticularly infiltrated, and which patients would benefit most from treatment, eliminating false expectations in the rest.

DETAILED DESCRIPTION:
This is the first clinical trial developed following the report of the Spanish Competent Authority on May 23, 2013, considering the PRP as a medicinal product for human use and establishing minimum guarantees required of the product and the process of manufacturing. It has been conducted from the perspective of both the trauma and the specialized treatment of chronic pain anesthesiologist, and manufacturing the PRP on the premises of a Regional Centre for Transfusions, all belonging to the Public Health System and therefore without commercial interests.

ELIGIBILITY:
Inclusion Criteria:

* Arthritis in the knee rated I, II, or III (Kellgren-Lawrence Grading Scale)
* VAS greater than 5
* Between 40and 80 years of age

Exclusion Criteria:

* Level IV arthritis of the knee
* Either surgery, corticoid infiltration, or viscosupplementation in the knee in the previous three months
* Frontal deformity greater than 10 degrees
* Ipsilateral pathology of the knee or ankle
* Range of motion or flexibility of the knee less than 90 degrees
* Deficit of knee extension greater than 15 degrees
* Anticoagulation treatment, antiplatelet treatment
* Hepatopathy
* Hematological neoplastic pathology
* Active infection
* Fibromyalgia
* Chronic fatigue syndrome

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Visual Analogue Scale (VAS) value | Evaluation will be conducted at 28 days,3 months and 6 months after first infiltration
  The main objective of this study is to determine the clinical value of intraarticular injections of platelet-rich plasma (PRP) in the reduction of perceived pain in patients with osteoarthritic knees

SECONDARY OUTCOMES:
Changes from baseline Knee and Osteoarthritis Outcome System (KOOS) scale value | Evaluation will be conducted at 28 days,3 months and 6 months after first infiltration
  KOOS is an instrument to assess the patient's opinion about their knee and associated problems. It includes 5 subscales which measure respectively the pain, symptoms, activities of daily living, sporting activity and quality of life
Effects on quality of life | Evaluation will be conducted at 28 days,3 months and 6 months after first infiltration
  EUROQOL (European Quality of Life) for the evaluation of function and quality of life
All reported adverse events | Evaluation will be conducted at 28 days,3 months and 6 months after first infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Montañez Heredia, MD, PhD, Principal Investigator — Hospital Universitario Virgen de la Victoria. Málaga